CLINICAL TRIAL: NCT06129188
Title: Comparison of Remimazolam With Propofol for Procedural Sedation in TEE
Brief Title: Comparison of Procedural Sedation in TEE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Justin Routman, MD, MSHA, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-300011945; UAB (Other: Anesthesiology)
Record Dates: First submitted 2023-10-31; First posted 2023-11-13 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Anesthesia
MeSH Terms: interventions — remimazolam; Propofol

STUDY DESIGN:
Intervention Model Description: After consenting to participate in the study, participants will undergo randomization in to one of two groups: those receiving remimazolam for sedation and those receiving propofol for sedation.
Who Masked: Participant
Masking Description: Of note, given the differences between propofol (premixed suspension, white color, weight-based dosing, often given via infusion, boluses typically vary from 3-10 mL doses) and remimazolam (requires reconstitution, clear color when reconstituted, non-weight-based dosing, only FDA approved for intermittent bolus administration, only FDA approved for boluses of 1-2 mL doses), it would not be possible for providers to be blinded to treatment group. Subjects and observers monitoring the MOAA/S level of sedation, however, will be blinded to treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Remimazolam (Experimental): 2.5-5 mg IV remimazolam will be administered no more frequently than every 2 minutes for the duration of the TEE procedure.
  Interventions: Drug: Remimazolam
- Propofol (Active Comparator): Standard-of-care IV propofol administration will be administered at the discretion of the anesthesia team caring for the patient for the duration of the TEE procedure
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam — Remimazolam is an ultra-short acting benzodiazepine medication. Benzodiazepines are a class of drug that directly interact with gamma-aminobutyric acid (GABA) and modifiable chloride channels through polysynaptic pathway inhibition. The anxiolytic properties of benzodiazepines make them useful as sedatives.
  Other Names: Byfavo
  Arms: Remimazolam
Drug: Propofol — Standard of care usage of the intravenous anesthetic agent propofol to achieve adequate sedation conditions for the procedure.
  Other Names: Diprivan
  Arms: Propofol

SUMMARY:
The objective of this proposal is to conduct a prospective randomized study comparing the utility of sedating patients undergoing transesophageal echocardiographic studies with a novel, recently-FDA-approved sedative agent, remimazolam, versus the sedative used in our current practice at UAB, propofol. This study will investigate whether remimazolam offers any benefit over current care vis-à-vis hemodynamics or efficiency/throughput.

This study will be conducted at the University of Alabama at Birmingham. All outpatients and inpatients scheduled for elective/non-emergent TEE in the UAB Heart and Vascular Center TEE lab will be considered for enrollment.

DETAILED DESCRIPTION:
Patients often undergo procedures outside of traditional operating rooms. With continued advances in minimally invasive and percutaneous techniques, recent trends demonstrate that sicker and increasingly unstable patients are routinely undergoing progressively more complex procedures in this space. Many of these procedures and patients necessitate varying levels of sedation due to pain, anxiety, and optimized procedural-conditions, among other reasons. Commonly utilized medications include benzodiazepines (like midazolam), opioids (like fentanyl), sedative-hypnotics (like propofol), and other adjuncts (such as dexmedetomidine and diphenhydramine).

Previous studies have shown that each of these agents has significant drawbacks that limit its utility. Propofol, while being fast in onset and offset, is limited by the lack of available reversal agent, the high liability for significant cardiac and/or respiratory depression, and the costly requirement of an anesthesia team for administration. Midazolam does not suffer from any of the shortcomings of propofol, but it has a much slower onset and offset, limiting both procedural and PACU timeliness/throughput and imparting prolonged CNS effects on patients (especially older patients) for hours to days after administration. Most adjuncts similarly have very slow onset and offset profiles, and they necessitate concomitant administration of other agents to achieve suitable procedural conditions.

Recently, a novel benzodiazepine (remimazolam) received FDA approval for procedural sedation for procedures lasting no more than thirty minutes. This agent combines the best qualities of propofol and midazolam while avoiding the downfalls of each. Specifically, remimazolam appears to maintain hemodynamic stability while rapidly allowing for ideal sedation conditions without lingering effects. These qualities make it a particularly good choice for procedural sedation and monitored anesthesia care for sicker, more tenuous patients. Despite FDA approval, adoption of this agent remains limited at present, likely due in part to cost as well as limited provider (anesthesiologist & proceduralist) experience with the agent. Nonetheless, it appears that using remimazolam for procedural sedation for our sickest patients with the most tenuous hemodynamic status may be a safer alternative to the current standard of care.

In attempt to answer this question, the investigators wish to compare the current practice of using propofol for sedation with the sedation achieved using remimazolam at recommended doses in patients scheduled to undergo transesophageal echocardiography. This patient population was intentionally chosen as it represents the sickest and most hemodynamically tenuous group of patients we sedate for procedures.

The significance of the study is that remimazolam, based on published experiences in other procedures, should produce robust sedation in subjects undergoing transesophageal echocardiogram studies with significantly less hemodynamic perturbation (hypotension) than results from propofol as part of current practice. If this observation is confirmed in this population, then it is likely that a change in the current practice would occur to improve patient safety.

Purpose: The purpose of this proposal is to conduct a prospective randomized study comparing the utility and safety of sedating patients for transesophageal echocardiographic studies with a novel, recently-FDA-approved sedative agent (remimazolam) versus the utility and safety of sedation produced by propofol.

Primary Hypothesis: Remimazolam will produce sedation for TEE procedures that is similar to that produced by propofol in terms of sedative conditions and speed of sedation onset/offset but will be associated with less hypotension.

Outline of Study:

The proposed study is a prospective randomized clinical study. All patients who undergo TEE already receive anesthesia care team-administered intravenous sedation during their procedures. In the present study, all groups will continue to receive standard-of-care treatment but will be randomized using a randomization generator to receive one of two different FDA-approved pharmacologic agents to achieve this sedation: remimazolam (a recently FDA-approved sedative hypnotic agent) and propofol (which is the agent most utilized in our practice). Baseline data collection in patients scheduled for elective/non-emergent inpatient or outpatient transesophageal echocardiogram will be collected. All physiologic variables (hemodynamic and respiratory parameters, body temperature, etc.) will be measured continually and recorded directly in the anesthesia procedure record. Similarly, all input/output data including any non-study medication administration (including but not limited to sedation and pressor agents), ongoing fluid, colloid and blood product administration will be recorded in the anesthesia record.

Assessment of the achieved level of sedation will be performed using the previously-validated Modified Observer's Assessment of Alertness/Sedation (MOAA/S) technique. Time to return to baseline neurologic status will be measured using the Modified Aldrete Scoring system as well as time from procedure finish to sign-out from the post anesthesia care unit by anesthesia providers.

Results from patients receiving remimazolam sedation will be compared to data from patients who receive propofol sedation. Since remimazolam will be new to the investigators' institution, there will be an option for the treating physician to convert their sedation plan from remimazolam to the more commonly utilized propofol if they do not feel the sedation is adequate. This will be an intention to treat (ITT) analysis.

Primary endpoints or outcomes: The primary endpoint will be the hemodynamic measures obtained throughout the transesophageal echocardiogram procedure. Secondary outcomes include a clinician assessment of the quality of the sedation, duration of onset of sedation, level of sedation, procedure duration, recovery duration, hemodynamic stability, required pressor use, complication rate, ICU stay, hospital stay, and 28- and 60-day mortality.

The investigators expect that patients will successfully be able to undergo a transesophageal echocardiogram using either remimazolam or propofol as a sole agent for sedation. The investigators expect that sedation conditions and speed of sedation onset and offset will be similar between the two groups. Most importantly, the investigators expect that there will be improved hemodynamic stability with use of remimazolam versus propofol (e.g., reduced hypotension and/or pressor requirement). The data collection, as proposed, should allow for all these comparisons in a statistically robust fashion.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients and outpatients >=18 years who are scheduled to undergo elective/non-emergent transesophageal echocardiography at the UAB Heart and Vascular Center TEE Lab.

Exclusion Criteria:

* Patients undergoing emergent TEE procedure in the HVC TEE Lab.
* Patients undergoing elective or emergent TEE procedure in the ICU and/or at the patient bedside.
* Patients undergoing elective or emergent TEE procedure in a location other than HVC TEE Lab.
* Patients undergoing an additional procedure or surgery (before or after TEE) as part of the same anesthetic, except for DC Cardioversion.
* Children under the age of 19 years (or under 50 kg body weight if age is unknown).
* Pregnant patients.
* Breastfeeding/nursing patients.
* Incarcerated patients.
* Patients enrolled in a concurrent ongoing interventional randomized clinical trial.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2025-02-25 (Actual); Primary Completion 2025-11-26 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Blood pressure, physiologic parameter | Only blood pressures recorded on the anesthesia record during the anesthetic administered for the TEE procedure.
  All patient blood pressure values (systolic and diastolic) recorded on the intraoperative anesthesia record.
Heart rate, physiologic parameter | Only heart rate recorded on the anesthesia record during the anesthetic administered for the TEE procedure.
  All patient heart rate values recorded on the intraoperative anesthesia record.

SECONDARY OUTCOMES:
Level of sedation, using the validated MOAA/S observer scale | Only values recorded during the TEE procedure
  Deepest level of sedation achieved during the TEE procedure as measured by an independent observer utilizing a validated scale. Scores range from 0-5, with 5 being fully awake and 0 being general anesthesia.
Duration of onset of sedation, using the validated MOAA/S observer scale | Only values recorded during the TEE procedure
  Duration of onset of sedation as measured from the time of medication administration until predetermined score on the scale is achieved, during the TEE procedure as measured by an independent observer utilizing a validated scale.Scores range from 0-5, with 5 being fully awake and 0 being general anesthesia.
Duration of procedure, recorded parameter | Only value recorded during the TEE procedure
  Total duration of the TEE procedure from probe insertion to removal, as recorded on the intraoperative anesthesia record.
Medication administration, recorded parameter | Only values recorded during the TEE procedure.
  All non-study medications administered during the TEE procedure will be recorded and aggregated. This information will be taken from the intraoperative anesthesia record. This will include the number of participants receiving any medication during the procedure other than the sedative to which they were randomized, what that medication was, what concentration dose was administered, the quantity of total doses were administered, and sum total dose administered per patient.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham Hospital, Birmingham, Alabama, United States